CLINICAL TRIAL: NCT07252466
Title: Factors Affecting Postnatal Mother-To-Infant Bonding: A Modelling Study
Brief Title: Factors Affecting Postnatal Mother-To-Infant Bonding
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assoc. Prof., Acibadem University
Other Study IDs: 62/2019
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Postpartum; Bonding; Newborn
Keywords: postnatal; bonding; infant; mothers-infant bonding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Term newborn-mother group: The group consists of mothers who gave birth at the hospital where the study was conducted during the data collection period and were found to be eligible to participate in the study, along with their infants. No intervention was performed on the mothers or infants.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was performed on the mothers or infants.

SUMMARY:
The aim of this study is to determine the factors that affect the postnatal mother-to-infant bonding.

DETAILED DESCRIPTION:
Bonding is recognised as one of the fundamental processes in terms of the socio-emotional development of the infants and the relationship they establish with the outside world.Mother-to-infant bonding typically initiates during pregnancy and continues to evolve through early childhood, reflecting the mother's emotional orientation toward her infant. The initial postnatal period is the most favourable time for the initiation of a positive mother-to-infant relationship and bonding.An adequate mother-to-infant bonding contributes to the positive physical and socio-emotional development of the child. A weaker mother-to-infant bonding is associated with insecure attachment and depression and anxiety in children. Also, women with weaker mother-to-infant bonding have been found to show less interest in the health of their children. These behaviours cause long-term negative cognitive and socio-emotional development in the child.In a study that assessed the level of mother-to-infant bonding in the postnatal period and the associated factors, in general, a significant proportion of mothers had difficulties in mother-to-infant bonding in the postnatal period. The postpartum period is a critical, complicated period of transition for both the mother and the infant, considering psychological, social, and physiological difficulties. Therefore, the mother-to-infant bonding can be affected by many factors. The aim of this study is to determine the factors that affect the postnatal mother-to-infant bonding.

ELIGIBILITY:
Inclusion Criteria:

* All healthy mothers who applied to the hospital's maternity ward at the time of the study
* who had a normal spontaneous delivery
* infants who were born at ≥38 gestational weeks
* infants who were deemed healthy by the physician were included in the study.

Exclusion Criteria:

* Mothers who had a risky health problem during delivery
* Infants who had a congenital illness

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mothers who give birth at the Maternity and Children's Hospital and their infants
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
MIBS level | Immediately after completion of the first breastfeeding
  After the first breastfeeding experience was completed, the mother assessed based on the mothers' self-reports using the Mother-Infant Bonding Scale (MIBS). The "MIBS", developed by Taylor et al., was used to assess mother-to-infant bonding following the first breastfeeding. The MIBS consists of 8 items rated on a 4-point Likert scale (0-3). Items 1, 4, and 6 assess positive emotions (scored as 0, 1, 2, 3), while items 2, 3, 5, 7, and 8 assess negative emotions (scored as 3, 2, 1, 0). Total scores range from 0 to 24, with lower scores indicating stronger mother-infant bonding. The tool has no specific cut-off value and has been shown to be sensitive in detecting subtle variations in early maternal bonding.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Coşkun, Assist.Prof., Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hailemeskel HS, Kebede AB, Fetene MT, Dagnaw FT. Mother-Infant Bonding and Its Associated Factors Among Mothers in the Postpartum Period, Northwest Ethiopia, 2021. Front Psychiatry. 2022 Jul 13;13:893505. doi: 10.3389/fpsyt.2022.893505. eCollection 2022. PMID 35911218
- [Result] Nakano M, Upadhyaya S, Chudal R, Skokauskas N, Luntamo T, Sourander A, Kaneko H. Risk factors for impaired maternal bonding when infants are 3 months old: a longitudinal population based study from Japan. BMC Psychiatry. 2019 Mar 8;19(1):87. doi: 10.1186/s12888-019-2068-9. PMID 30849963
- [Result] Ohara M, Okada T, Aleksic B, Morikawa M, Kubota C, Nakamura Y, Shiino T, Yamauchi A, Uno Y, Murase S, Goto S, Kanai A, Masuda T, Nakatochi M, Ando M, Ozaki N. Social support helps protect against perinatal bonding failure and depression among mothers: a prospective cohort study. Sci Rep. 2017 Aug 25;7(1):9546. doi: 10.1038/s41598-017-08768-3. PMID 28842556
- [Result] Taylor A, Atkins R, Kumar R, Adams D, Glover V. A new Mother-to-Infant Bonding Scale: links with early maternal mood. Arch Womens Ment Health. 2005 May;8(1):45-51. doi: 10.1007/s00737-005-0074-z. Epub 2005 May 4. PMID 15868385
- [Result] Tichelman E, Westerneng M, Witteveen AB, van Baar AL, van der Horst HE, de Jonge A, Berger MY, Schellevis FG, Burger H, Peters LL. Correlates of prenatal and postnatal mother-to-infant bonding quality: A systematic review. PLoS One. 2019 Sep 24;14(9):e0222998. doi: 10.1371/journal.pone.0222998. eCollection 2019. PMID 31550274